CLINICAL TRIAL: NCT00415038
Title: A Double Blind, Dose Range, Placebo Controlled Study of the Effects of Rostafuroxin vs Placebo in Patients With Stable, Uncomplicated, Essential Hypertension.
Brief Title: Efficacy of Rostafuroxin in the Treatment of Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Responsible Party: Giovanni Valentini, Sigma Tau i.f.r. S.p.A.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PST2238-DM-03-010
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Essential Hypertension
Keywords: hypertension; pharmacogenomic; adducin; ouabain; rostafuroxin
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — rostafuroxin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Rostafuroxin 50 micrograms capsules (Experimental): 5 weeks, once a day capsule treatment of active drug or placebo, followed by a 5 weeks, once a day capsule treatment of placebo or active drug according to a cross-over design
  Interventions: Drug: Rostafuroxin
- Rostafuroxin 150 micrograms capsules (Experimental): 5 weeks, once a day capsule treatment of active drug or placebo, followed by a 5 weeks, once a day capsule treatment of placebo or active drug according to a cross-over design
  Interventions: Drug: Rostafuroxin
- Rostafuroxin 500 micrograms capsules (Experimental): 5 weeks, once a day capsule treatment of active drug or placebo, followed by a 5 weeks, once a day capsule treatment of placebo or active drug according to a cross-over design
  Interventions: Drug: Rostafuroxin
- Rostafuroxin 1.5 mg capsules (Experimental): 5 weeks, once a day capsule treatment of active drug or placebo, followed by a 5 weeks, once a day capsule treatment of placebo or active drug according to a cross-over design
  Interventions: Drug: Rostafuroxin
- Rostafuroxin 5 mg capsule (Experimental): 5 weeks, once a day capsule treatment of active drug or placebo, followed by a 5 weeks, once a day capsule treatment of placebo or active drug according to a cross-over design
  Interventions: Drug: Rostafuroxin

INTERVENTIONS:
Drug: Rostafuroxin — 1 capusle of 50 micrograms of Rostafuroxin or placebo per day in the morning before breakfast for 5 weeks followed by other 5 weeks with placebo or Rostafuroxin
  Arms: Rostafuroxin 50 micrograms capsules
Drug: Rostafuroxin — 1 capusle of 150 micrograms of Rostafuroxin or placebo per day in the morning before breakfast for 5 weeks followed by other 5 weeks with placebo or Rostafuroxin
  Arms: Rostafuroxin 150 micrograms capsules
Drug: Rostafuroxin — 1 capusle of 500 micrograms of Rostafuroxin or placebo per day in the morning before breakfast for 5 weeks followed by other 5 weeks with placebo or Rostafuroxin
  Arms: Rostafuroxin 500 micrograms capsules
Drug: Rostafuroxin — 1 capusle of 1.5 milligrams of Rostafuroxin or placebo per day in the morning before breakfast for 5 weeks followed by other 5 weeks with placebo or Rostafuroxin
  Arms: Rostafuroxin 1.5 mg capsules
Drug: Rostafuroxin — 1 capusle of 5 milligrams of Rostafuroxin or placebo per day in the morning before breakfast for 5 weeks followed by other 5 weeks with placebo or Rostafuroxin
  Arms: Rostafuroxin 5 mg capsule

SUMMARY:
The purpose of this study is to verify the efficacy of Rostafuroxin in the treatment of essential hypertension and to determine the best effective dose to be administered in the general hypertensive population and in a subset of this population in which genetic patterns could be involved in the etiology of essential hypertension.

DETAILED DESCRIPTION:
Elevated arterial pressure is probably the most important public health problem. about 30% of the world adult population are affected by hypertension in industrialised countries. Development of a pharmacogenomic approach to the therapy of primary hypertension give new opportunities for the treatment of hypertension. This approach consists in the identification of the genetic-molecular mechanisms responsible for hypertension in a given subset of patients, and in the development of drugs able to interfere with such mechanisms, thus leading to very selective therapeutic interventions with enhanced efficacy and reduced side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade 1 or 2 of essential hypertension
* Less than 3 risk factors (age > 55 if male, smoking, dyslipidemia, family history of CV disease occurring before 55 years in men and 65 in women
* Naive patients or currently on monotherapy or one combination tablet
* SBP between 140 and 169 mmHg

Exclusion Criteria:

* Atrial fibrillation or left or right VBBB
* Left ventricular hypertrophy
* Significant renal or hepatic disease
* Obesity > 30kg/m2
* Diabetes mellitus

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 438 (Actual)
Dates: Start 2005-02; Primary Completion 2007-04 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Office Systolic Blood Pressure after 5 week of treatment | 5 weeks

SECONDARY OUTCOMES:
Office Diastolic Blood Pressure | 5 weeks
Proportion of normalised and responder patients (all visits) | 5 weeks
24 hours BP monitoring (through to peak ratio) | 5 weeks
Effect on sub-populations, genetically selected | 5 weeks
safety of the drug | monitored during all the study

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Staessen, MD PhD, Study Chair — Catholic University of Leuven, Laboratory of Hypertension Dept. of Molecular and cardiovascular Resesrach - Campus Gasthuisberg; Hilde Celis, MD, Principal Investigator — Catholic University of Leuven Dept. of Molecular and cardiovascular Research, Laboratory of Hypertension; Kalina Kawecka-Jaszcz, MD, Principal Investigator — Jagiellonian University Medical College Krakow - I Cardiac Department - Krakow (Poland); Bogdan Wyrzykowski, MD, Principal Investigator — Department of Hypertension and Diabetology - Medical Academy - Gdansk (Poland); Andrzej Tykarski, MD, Principal Investigator — Department of hypertension - School of Medicine - Poznan (Poland); Miroslaw Dluzniewski, MD, Principal Investigator — Postgraduate Medical School - Department of cardiology - Warszawa (Poland); Andrzey Januszewicz, MD, Principal Investigator — Department of Internal Medicine and Hypertension Warszawa (Poland); Tomasz Grodzicki, MD, Principal Investigator — Department of Internal Medicine and Gerontology - Jagiellonian University Medical College - Krakow (Poland); Wieslawa Piwowarska, MD, Principal Investigator — Coronary Disease Department - Jagiellonian University medical College - Krakow (Poland); Edoardo Casiglia, MD, Study Director — IV Clinica Medica dell'Università di Padova, Dipartimento di Medicina Clinica e Sperimentale - Padova (Italy); Giancarlo Basso, MD, Principal Investigator — U.O. Cardiologia - Ospedale Civile di Schio (Vicenza) Italy; Paolo Manunta, MD, Principal Investigator — Divisione di Nefrologia, Dialisi e Ipertensione - Ospedale S. Raffaele - Milano (Italy); Nicola Glorioso, MD, Principal Investigator — Centro per L'ipertensione A.S.L. n° 1 - Sassari (Italy); Gianni Bellomo, MD, Principal Investigator — Dipartimento di Medicina Interna, Nefrologia e dialisi - Ospedale San Giovanni Battista - Foligno (Perugia) Italy; Ezio Degli Esposti, MD, Principal Investigator — Unità di valutazione dell'efficacia clinica - Direzione Aziendale Ospedale S. Maria delle Croci - Ravenna (Italy); Yuri Nikitin, MD, Principal Investigator — Institute of internal Medicine, Siberian Branch of the Russian Academy of Medical Sciences - Novosibirsk (Russia); Viktor Milyagin, MD, Principal Investigator — Department of Internal Medicine, Postgraduate Education Faculty Smolensk State medical Academy - Smolensk (Russia); Sergey Nedogoda, MD, Principal Investigator — Department of Internal and family Medicine - Volgograd (Russia); James Barton, MD, Principal Investigator — Portiuncola Hospital Cardiac Research Department - Ballinasloe co Galway (Ireland); Peter W De Leeuw, MD, Principal Investigator — Academisch Ziekenhuis Maastricht Afdeling Nefrologie - Mastricht (The Netherlands); Marielle ME Krekels, MD, Principal Investigator — Department of Medicine/Nephrology Maaslandziekenhuis - Sittard (The Netherlands); Rock Accetto, MD, Principal Investigator — University Medical center, Hypertension Department - Ljubljana (Slovenia); Fernando Hernandez-Menarguez, MD, Principal Investigator — Centro de la Salud de Vistalegre - La Flota, Murcia (Spain); Jose a Aleman, MD, Principal Investigator — Centro de Salud Murcias San Andres - Murcia (Spain); Carlos c Gomez, MD, Principal Investigator — Hospital Clinico Universitario - Santiago de Compostela (Spain); Antonio Pose-Reino, MD, Principal Investigator — Hospital de Conxo - Santiago de Compostela (Spain); Jose M Pascual-Izuel, MD, Principal Investigator — Hospital de Sagunto - Sagunto (Valencia) - Spain; Josep Redon, MD, Principal Investigator — Hipertension Clinic, Hospital Clinico University of Valencia - Valencia (Spain); Antonio Coca-Payeras, MD, Principal Investigator — Hospital Clinico de Barcelona - Barcelona (Spain); Jan Filipovsky, MD, Principal Investigator — Derpartment of Internal Medicine 2, Faculty of Medicine - Pilsen (Czech Republic); Miroslav Soucek, MD, Principal Investigator — Department of Internal Medicine 2, St. Anne's Hospital, Faculty of Medicine - Brno (Czech Republic); Michel Burnier, MD, Principal Investigator — Division de Nephrologie, Department de Medecine, Centre Hopitalier Universitaire Vaudois - Lausanne (Switzerland)
Locations (1):
- Catholic University of Leuven - Laboratory of Hypertension, Dept. of Molecular and Cardiov. Research - Campus Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Background] Staessen JA, Kuznetsova T, Acceto R, Bacchieri A, Brand E, Burnier M, Celis H, Citterio L, de Leeuw PW, Filipovsky J, Fournier A, Kawecka-Jaszcz K, Manunta P, Nikitin Y, O'Brien ET, Redon J, Thijs L, Ferrari P, Valentini G, Bianchi G. OASIS-HT: design of a pharmacogenomic dose-finding study. Pharmacogenomics. 2005 Oct;6(7):755-75. doi: 10.2217/14622416.6.7.755. PMID 16207152
- [Derived] Staessen JA, Thijs L, Stolarz-Skrzypek K, Bacchieri A, Barton J, Espositi ED, de Leeuw PW, Dluzniewski M, Glorioso N, Januszewicz A, Manunta P, Milyagin V, Nikitin Y, Soucek M, Lanzani C, Citterio L, Timio M, Tykarski A, Ferrari P, Valentini G, Kawecka-Jaszcz K, Bianchi G. Main results of the ouabain and adducin for Specific Intervention on Sodium in Hypertension Trial (OASIS-HT): a randomized placebo-controlled phase-2 dose-finding study of rostafuroxin. Trials. 2011 Jan 14;12:13. doi: 10.1186/1745-6215-12-13. PMID 21235787